CLINICAL TRIAL: NCT04972123
Title: The Effect of Capsaicin-Phenylephrine-Caffeine Formulation on Aborting Tilt Induced Syncope in Patients With a History of Vasovagal Syncope or Near Syncope
Brief Title: The Effect of CPC on Aborting Tilt Induced Syncope in Patients With a History of Vasovagal Syncope or Near Syncope
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2021-0081; Protocol Version 4/12/2022 (Other: UW Madison); A534225 (Other: UW Madison); SMPH/MEDICINE/CARDIOLOGY (Other: UW Madison)
Record Dates: First submitted 2021-07-12; First posted 2021-07-22 (Actual); Results first posted 2024-06-24 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-06

CONDITIONS: Syncope, Vasovagal
Keywords: Neurocardiogenic Syncope; Reflex Syncope; Fainting Spells
MeSH Terms: conditions — Syncope, Vasovagal; Syncope | interventions — Phenylephrine; Caffeine; Tilt-Table Test

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Randomized 1:1 to CPC or placebo
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CPC Adminstration (Experimental): Single dose of CPC will be given during tilt table test
  Interventions: Drug: CPC - Capsaicin, Phenylephrine, Caffeine; Diagnostic Test: Tilt Table Test
- Placebo Adminstration (Placebo Comparator): Single dose of Placebo will be given during tilt table test
  Interventions: Diagnostic Test: Tilt Table Test; Drug: Placebo

INTERVENTIONS:
Drug: CPC - Capsaicin, Phenylephrine, Caffeine — CPC is a combination of Capsaicin, Phenylephrine and Caffeine
  Arms: CPC Adminstration
Diagnostic Test: Tilt Table Test — Participant will undergo tilt tablet testing using the Italian protocol (see reference section). The Italian protocol includes 20 minutes of passive tilt at 70 degrees (Passive Phase) followed by nitroglycerin (NTG) administration and tilt testing for another 15 minutes (NTG Phase).
Drug: Placebo — Placebo for CPC
  Arms: Placebo Adminstration

SUMMARY:
Syncope is defined as transient loss of consciousness associated with inability to maintain postural tone with rapid and spontaneous recovery. The purpose of this study is to assess the effects of sublingual administration of a new medication called CPC on tilt-induced syncope in patients with a history of vasovagal syncope (VVS) or near syncope. 140 participants will be randomized at the University of Wisconsin - Madison. Each participant will be in the study for 1 day.

DETAILED DESCRIPTION:
Vasovagal syncope (VVS) is the most common type of syncope. The mechanism is reflex-mediated triggered by various afferent input to the brain. The event is usually preceded by diaphoresis, warmth, nausea, and pallor, and is followed by fatigue. While several drugs are indicated in the treatment of VVS, to our knowledge, there is no current treatment of an impending syncopal attack. In the present study, the investigators hypothesized that a single administration of sublingual CPC preparation during the prodromal phase would abort tilt-induced syncope or near syncope with SBP less than or equal to 70 mmHg in patients with a history of VVS. Patients with an established diagnosis of typical VVS or near syncope will be randomized to receive CPC or placebo in 1:1 ratio. Drug or placebo will be administered at the onset of prodromes during tilt table testing. In addition to the primary endpoint (syncope or near syncope with SBP less than or equal to 70 mmHg), the investigators will be assessing the effects of the drug on time to event, incidence of asystole (> 3 sec), and fatigue after syncope.

ELIGIBILITY:
Inclusion Criteria:

1. Established diagnosis of typical vasovagal syncope or near syncope
2. Age 18-50 years

Exclusion Criteria:

1. Systolic BP >130 mmHg
2. History of hypertension or cardiac arrhythmias
3. History of cardiovascular disease or cerebral ischemic events
4. Allergic reaction to any of the drug components
5. Contraindication to tilt testing
6. Any physical or psychological symptom, based on the clinical judgment of the investigators that would make a participant unsuitable for the study
7. Any use of a medication(s) based on the clinical judgment of the investigators that would make a participant unsuitable for the study (e.g. fludrocortisone, theophylline, prazosin, doxazosin, terazosin, MAO-inhibitors, pseudoephedrine, decongestant and PDE5 inhibitors).
8. Unwilling to discontinue Midodrine or beta-blocker therapy 48 hours before tilt table testing.
9. Women who are pregnant (confirmed with pregnancy test on day of study) or lactating.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 143 (Actual)
Dates: Start 2021-07-20 (Actual); Primary Completion 2023-08-25 (Actual); Study Completion 2023-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed H Hamdan, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin- Madsion, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bartoletti A, Alboni P, Ammirati F, Brignole M, Del Rosso A, Foglia Manzillo G, Menozzi C, Raviele A, Sutton R. 'The Italian Protocol': a simplified head-up tilt testing potentiated with oral nitroglycerin to assess patients with unexplained syncope. Europace. 2000 Oct;2(4):339-42. doi: 10.1053/eupc.2000.0125. PMID 11194602

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at the University of Wisconsin- Madison using general recruitment emails addressed to students, faculty and staff and UW Heath Faint and Fall Clinic patients. All participants signed electronic consents in advance of study visit. The first participant completed the study in July 2021, and the last participant completed the study in August 2023.
Pre-assignment Details: Digital consent was obtained in 143 subjects. 14 subjects were not randomized for various reasons; no show (n=3), withdrew consent (n=4), SBP > 130 mmHg (n=6) and not withholding Midodrine (n=1). A total of 129 subjects were randomized to CPC (n=66) or Placebo (n=63).
Groups:
- CPC Adminstration: Single dose of CPC will be given during tilt table test at onset of prodromes. CPC - Capsaicin, Phenylephrine, Caffeine
- Placebo Adminstration: Single dose of Placebo will be given during tilt table test at onset of prodromes
Period: Overall Study
Arm/Group | CPC Adminstration | Placebo Adminstration
Started | 66 | 63
Primary Analysis Population (Primary Analysis was completed for participants where BP could be obtained at the time of near syncope (technical issues for N=2 participants where BP could not be obtained)) | 65 | 62
Secondary Analysis Population (Secondary analyses were limited to participants who had syncope or near syncope with systolic BP less than or equal to 70 mmHg) | 32 | 27
Completed | 66 | 63
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Evaluable participants for intention to treat primary endpoint By protocol entry criteria the age range was 18 to 50 Years.
Groups:
- CPC Adminstration: Participant who were randomized to received CPC during Tilt Testing for which evaluable data was available.
- Placebo Administration: Participant who were randomized to received Placebo during Tilt Testing for which evaluable data was available.
- Total: Total of all reporting groups
Arm/Group | CPC Adminstration | Placebo Administration | Total
Number analyzed (Participants) | 65 | 62 | 127
Age, Continuous [Median (Standard Deviation); unit: Years] | 26.2 (7.1) | 26.2 (7.5) | 26.2 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 55 | 110
  Male | 10 | 7 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 2 | 6
  Not Hispanic or Latino | 54 | 55 | 109
  Unknown or Not Reported | 7 | 5 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 5 | 6 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 0 | 3
  White | 48 | 47 | 95
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 8 | 9 | 17
Region of Enrollment [Number; unit: participants]
  United States | 65 | 62 | 127
Syncope History [Count of Participants; unit: Participants] — Participants who have a health history of Syncope or Near Syncope.
  Participants
    Participants with a history of syncope | 60 | 58 | 118
    Participant with a history of near syncope | 5 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Have Hypotensive Syncope or Near Syncope With SBP Less Than or Equal to 70 mmHG During Tilt Test
Description: Hypotensive syncope is defined as transient loss of consciousness associated with SBP less than or equal to 90 mmHg. Near syncope is defined as sensation of "near fainting" while still being responsive to verbal commands. Near syncope will be used as a primary endpoint only when it is associated with a SBP less than or equal to 70 mmHg.
Time Frame: During tilt table testing (up to approximately 35 minutes)
Population: Intention to treat based on randomized treatment assignment
Measure: Count of Participants; unit: Participants
Arm/Group | CPC Adminstration | Placebo Administration
Number analyzed (Participants) | 65 | 62
Participants
  Number of participants with syncope or near syncope event | 32 | 27
  Number of participants without syncope or near syncope event | 33 | 35
Statistical Analysis 1: Comparison: CPC Adminstration vs Placebo Administration; Primary endpoint -- ITT primary endpoint analysis; Test type: Superiority — The primary end point was evaluated via a large sample Z-test for proportions. The test statistic was compared to a Pocock monitoring boundary at both an interim analysis and at the final analysis; p = 0.521, Large sample Z-test for population prop — The primary end point was evaluated via a large sample Z-test for proportions. The test statistic was compared to a Pocock monitoring boundary at both an interim analysis and at the final analysis; The test statistic was compared to a Pocock monitoring boundary at both an interim analysis and at the final analysis

2. Primary Outcome: Time to Syncope or Near-syncope After CPC or Placebo Administration
Description: Time in seconds from CPC or Placebo administration to syncope or near syncope in patients who had an event
Time Frame: During tilt table testing (up to approximately 35 minutes)
Population: Secondary endpoints analyses were limited to participants who had syncope or near syncope
Measure: Median (Standard Deviation); unit: seconds
Groups:
- CPC Administration: Participants randomized to receive CPC who experienced an event
- Placebo Administration: Participants randomized to receive Placebo who experienced an event
Arm/Group | CPC Administration | Placebo Administration
Number analyzed (Participants) | 32 | 27
seconds | 90.1 (95.0) | 76.9 (95.0)
Statistical Analysis 1: Comparison: CPC Administration vs Placebo Administration; Secondary endpoint -- Time to event for evaluable ITT population who had a primary event; Test type: Superiority — Time to event was compared between groups via a log-rank test; p = 0.574, Log Rank — Time to event was compared between groups via a log-rank test

3. Secondary Outcome: Percentage of Patients Who Have Asystolic Pauses > 3 Seconds in the CPC and Placebo Arms
Description: Percentage of Participants with an event who had asystolic pauses > 3 seconds during syncope or near syncope
Time Frame: During tilt table testing (up to approximately 35 minutes)
Population: Secondary endpoints analyses were limited to participants who had syncope or near syncope
Measure: Count of Participants; unit: Participants
Arm/Group | CPC Administration | Placebo Administration
Number analyzed (Participants) | 32 | 27
Participants | 2 | 1
Statistical Analysis 1: Comparison: CPC Administration vs Placebo Administration; Secondary endpoint -- Incidence of asystolic pause > 3 seconds for evaluable ITT population who had a primary event; Test type: Superiority — Incidence of asystole were compared between groups using Fisher exact test; p = 1.000, Fisher Exact — Incidence of asystole were compared between groups using Fisher exact test; Incidence of asystole were compared between groups using Fisher exact test

4. Secondary Outcome: Fatigue Scores at 1, 4, and 8 Hours Post Tilt Table Testing
Description: Fatigue Scores at 1, 4 and 8 hours post tilt table testing in participants who had an event. Using standard continuous fatigue scale of 1 to 5, with 1 = no fatigue and 5 = max fatigue.
Time Frame: Up to 8 hours after tilt table testing (up to approximately 8 hours and 35 minutes)
Population: Secondary endpoints analyses were limited to participants who had syncope or near syncope
Measure: Median (Standard Deviation); unit: Score on a scale
Groups:
- CPC Adminstration: Participants randomized to receive CPC who experienced an event
Arm/Group | CPC Adminstration | Placebo Administration
Number analyzed (Participants) | 32 | 27
Score on a scale
  Fatigue rated at 1 hour post tilt test | 2.2 (1.05) | 2.0 (0.85)
  Fatigue rated at 4 hour post tilt test | 2.2 (1.09) | 2.3 (1.07)
  Fatigue rated at 8 hour post tilt test | 1.9 (0.91) | 2.6 (1.39)
Statistical Analysis 1: Comparison: CPC Adminstration vs Placebo Administration; Secondary endpoint -- Measures of Fatigue for evaluable ITT population who had a primary event; Test type: Superiority — Reporting for the 1 hour fatigue score only; p = 0.732, Wilcoxon (Mann-Whitney) — Measures of fatigue were compared between groups using the Wilcoxon rank-sum test; Measures of fatigue were compared between groups using the Wilcoxon rank-sum test
Statistical Analysis 2: Comparison: CPC Adminstration vs Placebo Administration; Secondary endpoint -- Measures of Fatigue for evaluable ITT population who had a primary event; Test type: Superiority — Reporting for the 4 hour fatigue score only; p = 0.591, Wilcoxon (Mann-Whitney) — Measures of fatigue were compared between groups using the Wilcoxon rank-sum test; Measures of fatigue were compared between groups using the Wilcoxon rank-sum test
Statistical Analysis 3: Comparison: CPC Adminstration vs Placebo Administration; Secondary endpoint -- Measures of Fatigue for evaluable ITT population who had a primary event; Test type: Superiority — Reporting for the 8 hour fatigue score only; p = 0.034, Wilcoxon (Mann-Whitney) — Measures of fatigue were compared between groups using the Wilcoxon rank-sum test; Measures of fatigue were compared between groups using the Wilcoxon rank-sum test

ADVERSE EVENTS:
Time Frame: Start of study visit to 8 hours post CPC or Placebo administration
Description: All symptoms reported by a participant that were unexpected in terms of intensity or duration were reported even if no study medication was given. The signs and symptoms associated with prodromes or events i.e. vasovagal syncope or near syncope were not reported as adverse events.
Groups:
- CPC Adminstration: Participants who were randomized to received CPC during Tilt Testing
- Placebo Administration: Participants who were randomized to received Placebo during Tilt Testing
Arm/Group | CPC Adminstration | Placebo Administration
All-Cause Mortality (participants affected / at risk) | 0/66 | 0/63
Serious Adverse Events (participants affected / at risk) | 0/66 | 0/63
Other Adverse Events (participants affected / at risk) | 3/66 | 4/63
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CPC Adminstration (N=66) | Placebo Administration (N=63)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 3 (3)
Migraine Headache (Nervous system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-05-04): https://cdn.clinicaltrials.gov/large-docs/23/NCT04972123/Prot_SAP_000.pdf
  • Informed Consent Form (2023-05-23): https://cdn.clinicaltrials.gov/large-docs/23/NCT04972123/ICF_001.pdf